CLINICAL TRIAL: NCT04942821
Title: Treatment of Multiple Adjacent Gingival Recessions With Coronally Advanced Flap in Combination With Platelet-Rich Fibrin: A Split-Mouth Study
Brief Title: The Evaluation Clinical Results of Coronally Advanced Flap With Platelet Rich Fibrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-04-2014/418
Record Dates: First submitted 2021-06-07; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2019-03

CONDITIONS: Root Coverage
Keywords: Gingival recession; Plastic surgery; Platelet rich fibrin; Connective tissue graft; Coronally advanced flap
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich fibrin and coronally advanced flap (Experimental): Coronally advanced flap and platelet rich fibrin were used in treatment arms.
  Interventions: Procedure: Platelet rich fibrin and coronally advanced flap
- Connective tissue graft and coronally advanced flap (Active Comparator): Coronally advanced flap and connective tissue graft were used in treatment arms.
  Interventions: Procedure: Connective tissue graft and coronally advanced flap

INTERVENTIONS:
Procedure: Platelet rich fibrin and coronally advanced flap — CAF were used in treatment arms. Root planning was performed on the exposed part of roots to provide more biocompatible surface for re-attachment. Two 10 cc tubes with clot activator were used to collect blood from the patient; blood was centrifuged at 2700 rpm for 12 min. PRF box was used to form fibrin clots into membranes. PRF was positioned at the level of the cemento-enamel junction (CEJ), and sutured on the periosteum bed with 6/0 absorbable sutures. Gingival margins on the flap were placed at least 1 mm coronally of the CEJ and sutured with 5/0 absorbable sutures. Sutures were removed at 2nd week.
  Arms: Platelet rich fibrin and coronally advanced flap
Procedure: Connective tissue graft and coronally advanced flap — Control sites were treated by coronally advanced flap (CAF) combined with connective tissue graft (CTG). CAF were used in both treatment arms. Root planning was performed on the exposed part of roots to provide more biocompatible surface for re-attachment. CTG was obtained with single incision method. CTG was positioned at the level of the cemento-enamel junction (CEJ), and sutured on the periosteum bed with 6/0 absorbable sutures. Gingival margins on the flap were placed at least 1 mm coronally of the CEJ and sutured with 5/0 absorbable sutures. Sutures were removed at 2nd week.
  Arms: Connective tissue graft and coronally advanced flap

SUMMARY:
The aim of this study was to evaluate the clinical outcomes of platelet- rich fibrin and coronally advanced flap technique in the treatment of multiple gingival recessions in comparison with connective tissue graft technique.

DETAILED DESCRIPTION:
Aim of this study was to evaluate the clinical outcomes of platelet rich fibrin (PRF)+coronally advanced flap (CAF) technique in the treatment of multiple gingival recessions in comparison with connective tissue graft (CTG)+CAF technique.12 patients with bilateral Miller Class I multiple gingival recessions were treated with PRF+CAF (test group) and CTG+CAF (control group) technique in a split-mouth study design. Probing depth, recession depth (RD), clinical attachment level (CAL), recession width, position of gingival margin, papilla width, keratinized tissue height (KTH), keratinized tissue thickness (KTT) were measured at baseline and 3, 6 and 12 months after surgery. Root coverage (RC) and complete root coverage (CRC) ratios were evaluated post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients had at two quadrants, adjacent Miller Class I and at least 2 mm or deeper recessions
* Full mouth plaque score 20% and Full mouth bleeding on probing 10%
* no active periodontal disease,
* involving incisors, canines and premolars,
* age ≥ 18 years

Exclusion Criteria:

* Patients with general diseases which could affect healing process,
* smokers
* Patients had undergone periodontal surgery during the pervious 24 months on the involved sites,
* pregnant or breastfeeding women
* endodontic lesions or non-detectable cemento-enamel junctions at experimental teeth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04-23 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Root Coverage | 12 months
  The percentage of root coverage was calculated according to the preoperative recession depth to postoperative recession depth.

SECONDARY OUTCOMES:
Complete Root Coverage | 12 months
  Complete root coverage was calculated according to measurement of the pre and post operative gingival margin which was above the enamel-sement junction.
Change from Baseline Keratinized Tissue Width at 3 months | 3 months
  Width of keratinized tissue at mid-buccal point measured from free gingival margin to mucogingival junction
Change from Baseline Keratinized Tissue Width at 6 months | 6 months
  Width of keratinized tissue at mid-buccal point measured from free gingival margin to mucogingival junction
Change from Baseline Keratinized Tissue Width at 12 months | 12 months
  Width of keratinized tissue at mid-buccal point measured from free gingival margin to mucogingival junction
Change from Baseline Gingival Thickness at 3 months | 3 months
  Gingival thickness at mid-buccal aspect measured at the center of keratinized tissue.
Change from Baseline Gingival Thickness at 6 months | 6 months
  Gingival thickness at mid-buccal aspect measured at the center of keratinized tissue.
Change from Baseline Gingival Thickness at 12 months | 12 months
  Gingival thickness at mid-buccal aspect measured at the center of keratinized tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Selin Yıldırım, Dr., Study Chair — Marmara University, Faculty of Denistry, Department of Periodontology; Başak Doğan, Prof. Dr., Study Director — Marmara University, Faculty of Denistry, Department of Periodontology; Atacan Yavuz, Dr., Principal Investigator — Marmara University, Faculty of Denistry, Department of Periodontology

REFERENCES:
- [Derived] Yavuz A, Gungormek HS, Kuru L, Dogan B. Treatment of multiple adjacent gingival recessions using leucocyte- and platelet-rich fibrin with coronally advanced flap: a 12-month split-mouth controlled randomized clinical trial. Clin Oral Investig. 2024 May 1;28(5):291. doi: 10.1007/s00784-024-05694-3. PMID 38691209